CLINICAL TRIAL: NCT06583460
Title: Systematic Intervention to Improve Sexual Dysfunction in Adjuvant Breast Cancer Patients
Brief Title: Systematic Intervention to Improve Sexual Dysfunction
Acronym: SISTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-4-72-002; 2023-A02035-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-08-06; First posted 2024-09-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Female; Localized Cancer
Keywords: Sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Category 2 clinical trial, monocentric, prospective, comparative, controlled but not randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer treatment with oncosexology supporting care (Other): Patient initially treated by surgery combined with any therapy (chemotherapy, radiotherapy, hormonal therapy etc.) and benefiting oncosexological care.
  Interventions: Other: Early and systematic oncosexological supporting care

INTERVENTIONS:
Other: Early and systematic oncosexological supporting care — Each patient included in the study will be cared by an anthropologist and a sexologist.
  This therapeutic support care will be based on :
  * 2 qualitative semi-directive interviews (Baseline and M18),
  * 2 individual consultations with questionnaires (Baseline and M18).
  The qualitative semi-structured interviews will be conducted with the anthropologist, and the individual consultations with the sexologist.
  At the end of the first oncosexology consultation, patients will be given the opportunity to decide whether or not to accept further systematic oncosexology support care, which will be based on :
  * 3 individual and/or couple consultations,
  * 3 group workshops.
  Patients are under no obligation to accept this additional oncosexology support care.

SUMMARY:
The aim of this clinical trial is to compare the benefit of early, systematic, multidisciplinary oncosexological care versus on-demand care on the sexual health of women with breast cancer.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of early, systematized oncosexology care on perceived sexual health at 18 months, compared with oncosexology care on demand.

All included patients are evaluated at Baseline and M18 following initiation of antineoplastic treatments associated with surgery. Patients who accepted additional oncosexological care were also assessed at M4, M8 and M12. The content of support care is detailed in section "arms and interventions".

Oncosexology consultations with the sexologist and the medical support care of any organic disorders remain accessible to all patients, on request, including the group of patients who do not wish to participate in early and systematic oncosexology care.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years (menopausal or not),
* Localized breast cancer with or without lymph node involvement,
* Initial treatment starting with surgical resection, whatever the associated therapy (chemotherapy, radiotherapy, hormone therapy, monoclonal antibody, conjugated drug antibody, targeted therapy such as cyclin and anti-PARP inhibitors, etc.),
* Patient affiliated or benefiting from the social security system,
* Patient informed and informed consent signed.

Exclusion Criteria:

* History of cancer (except squamous cell carcinoma or basal cell carcinoma) in the last five years,
* Pregnant or breast-feeding women,
* Patients deprived of their liberty, under guardianship or curatorship and all other administrative safeguards,
* Patients unable to comply with the study schedule for social, medical or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-06-09 (Estimated); Study Completion 2028-06-09 (Estimated)

PRIMARY OUTCOMES:
Sexual satisfaction | Measured at baseline and at 18 months following initiation of treatment and surgical.
  Sexual satisfaction score measured by self-questionnaire using the EORTC Quality of Life Questionnaire Sexual Health scale (EORTC QLQ-SH22).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lefeuvre-Plesse, MD, Principal Investigator — Centre de Lutte Contre Le cancer Eugène Marquis
Locations (1):
- Centre de Lutte contre le Cancer Eugène Marquis, Rennes, Brittany Region, France